CLINICAL TRIAL: NCT00203814
Title: Open-Label, Randomised, Parallel Group in Vivo Drug Study to Evaluate Combination Anti-Malarial Therapy (CAT), Artesunate and Sulfadoxine-Pyrimethamine Versus Sulfadoxine-Pyrimethamine Alone, in Terms of Therapeutic Efficacy, Prevalence of Gametocyte Carriage and Prevalence of Molecular Markers Associated With SP Resistance In Uncomplicated Plasmodium Falciparum Infections.
Brief Title: A Randomised Efficacy Study of Combination Antimalarials to Treat Uncomplicated Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: World Health Organization (Other); Medical Research Council, South Africa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEACAT 01a ASSP
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2005-08

CONDITIONS: Malaria
Keywords: Malaria; Efficacy; Pharmacokinetic; Gametocyte; Molecular markers; Sulfadoxine-pyrimethamine; Artesunate; Artemisinin
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Artesunate

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine
Drug: Artesunate plus sulfadoxine-pyrimethamine

SUMMARY:
The purpose of this study is to determine the efficacy of sulfadoxine-pyrimethamine plus artesunate versus sulfadoxine-pyrimethamine alone in the treatment of uncomplicated malaria.

DETAILED DESCRIPTION:
Resistance of Plasmodium falciparum to anti-malarial drugs is a serious impediment to the control of malaria. In order to facilitate formulation of effective regional drug policies and to provide a database for decision-making on the implementation of combination therapy (CAT), it is essential that the in vivo response to CAT be investigated. In the South East African Combination Anti-malarial Therapy (SEACAT) evaluation, there is a comprehensive evaluation of the phased introduction of combination anti-malarial therapy in Mozambique. As a component of this evaluation, in selected Mozambique sites where intensity of malaria transmission is high, a direct parallel group comparison of monotherapy (SP) with CAT (artesunate plus SP) will be conducted according to this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, older than 12 months.
* Weight > 10 kg.
* Diagnoses of pure uncomplicated acute P. falciparum malaria parasitaemia of up to 500 000 asexual parasite/mcl blood with axillary temperature of greater than or equal to 37.5°C or history of fever (defined as within the previous 24 hours).
* Documented informed consent.
* Lives close enough to the study site for reliable follow up.

Exclusion Criteria:

* Has received anti-malarial treatment in the past 7 days.
* Is infected with other malarial species (such subjects may be excluded retrospectively from the analysis).
* Severely ill (based on WHO Criteria for severe malaria ) or if patient is considered, in the opinion of the investigator or designee, to have moderately severe malaria (e.g. prostrate, repeated vomiting, dehydrated) or other danger signs.
* Has received cotrimoxazole, trimethoprim, chloramphenicol, folate or tetracyclines (including doxycycline) in the past 7 days or is likely to require these during the study period.
* History of G6PD deficiency.
* Is pregnant or breastfeeding.
* Has a history of allergy to any of the study drugs (including other sulphonamides e.g. cotrimoxazole, other artemisinin derivatives e.g. co-artemether).
* Serious underlying disease that in the opinion of the clinic team and/or Principal Investigator would make the patient unsuitable for the study in terms of their safety or study analysis.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280
Dates: Start 2004-01; Study Completion 2005-03

PRIMARY OUTCOMES:
Therapeutic efficacy defined as:Adequate Clinical and Parasitological Response (ACPR), Early Treatment Failure (ETF), Late Treatment Failure (LTF), defined as Late Clinical Failure (LCF) and Late Parasitological Failure (LPF)
Sensitive or parasitological failure (RI, early and late, RII, RIII)
Parasitological failures will be classified as recrudescence or re-infection (or indeterminate) using GLURP and MSP I & II markers
Parasite clearance time
Fever clearance time

SECONDARY OUTCOMES:
Association between study treatment and gametocyte carriage
Pharmacokinetics by measurement of whole blood levels of Sulfadoxine and Pyrimethamine
Correlation of the frequency of DHFR and DHPS mutations with parasitological outcome
Tolerability by describing adverse events and changes in haematological parameters
Capacity building by describing the training and development of study teams and their subsequent skills attained

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barnes, MBChB, Principal Investigator — University of Cape Town
Locations (2):
- Mozambique (2):
  - Boane Clinic, Boane, Maputo Province
  - Magude Clinic, Magude

REFERENCES:
- [Derived] Allen EN, Little F, Camba T, Cassam Y, Raman J, Boulle A, Barnes KI. Efficacy of sulphadoxine-pyrimethamine with or without artesunate for the treatment of uncomplicated Plasmodium falciparum malaria in southern Mozambique: a randomized controlled trial. Malar J. 2009 Jun 26;8:141. doi: 10.1186/1475-2875-8-141. PMID 19558654